CLINICAL TRIAL: NCT00003432
Title: A Phase I/II Study of Active Immunotherapy With Carcinoembryonic Antigen RNA-Pulsed, Autologous Cultured Dendritic Cells for Patients With Breast Cancer Who Achieve a Complete Response After High Dose Chemotherapy and Stem Cell Support
Brief Title: Immunotherapy in Treating Patients With Metastatic Breast Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: low accrual
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2030; IRB 2030 (Other: DUMC); CDR0000066458 (Other: NCI)
Record Dates: First submitted 1999-11-01; First posted 2003-04-25 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2013-11

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- carcinoembryonic antigen RNA-pulsed DC cancer vaccine (Experimental): carcinoembryonic antigen RNA-pulsed DC cancer vaccine
  Interventions: Biological: carcinoembryonic antigen RNA-pulsed DC cancer vaccine

INTERVENTIONS:
Biological: carcinoembryonic antigen RNA-pulsed DC cancer vaccine — Approximately 60-90 days after the peripheral blood stem cell transplant, patients receive CEA RNA pulsed dendritic cells IV every 3 weeks for a total of 4 doses.

SUMMARY:
RATIONALE: Immunotherapy using CEA-treated white blood cells may help a person's body build an immune response to and kill their tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of immunotherapy with CEA-treated white blood cells in treating patients with metastatic breast cancer who have achieved a partial or complete response after chemotherapy and peripheral stem cell transplantation.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the ability of active immunotherapy with carcinoembryonic antigen (CEA) RNA pulsed dendritic cells to induce CEA specific T cells in patients with metastatic breast cancer in complete remission following peripheral blood stem cell transplant.
* Determine the clinical efficacy in terms of overall and recurrence free survival of immunotherapy with CEA RNA pulsed dendritic cells in this patients population.

OUTLINE: Dendritic cells are taken from the leukapheresis product obtained during the peripheral blood stem cell transplant procedure performed prior to treatment on this study. The dendritic cells are pulsed with carcinoembryonic antigen (CEA) RNA. Approximately 60-90 days after the peripheral blood stem cell transplant, patients receive CEA RNA pulsed dendritic cells IV every 3 weeks for a total of 4 doses. Patients undergo a second leukopheresis after the last dose of immunotherapy to obtain specimens for immunologic tests.

Patients are followed every 3 months for the first year and annually thereafter.

PROJECTED ACCRUAL: A total of 14-26 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic breast cancer that expresses carcinoembryonic antigen (CEA)

  * At least 25% of the tumor cells must stain positive for CEA with at least moderate intensity
* Must have achieved either partial response or complete response after high dose chemotherapy and peripheral blood stem cell transplant
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Menopausal status:

* Not specified

Performance status:

* Karnofsky 70-100%

Life expectancy:

* Greater than 6 months

Hematopoietic:

* Absolute neutrophil count at least 1000/mm^3
* Absolute lymphocyte count at least 1000/mm^3
* Hemoglobin at least 9 mg/dL
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin less than 2.0 mg/dL
* No serious ongoing chronic or acute hepatic disease

Renal:

* Creatinine less than 2.5 mg/dL

Cardiovascular:

* No serious ongoing chronic or acute cardiac disease (New York Heart Association class III or IV)

Pulmonary:

* No serious ongoing chronic or acute pulmonary illness such as asthma, chronic obstructive pulmonary disease, or radiation or drug induced pneumonitis

Other:

* No other prior or concurrent malignancy except nonmelanoma skin cancer or controlled superficial bladder cancer within the past 5 years
* No history of autoimmune disease such as inflammatory bowel disease, systemic lupus erythematosus, rheumatoid arthritis, ankylosing spondylitis, scleroderma, or multiple sclerosis
* No inflammatory bowel condition such as active infectious enteritis or eosinophilic enteritis
* No active acute or chronic infection such as urinary tract infection, HIV, or viral hepatitis
* Not pregnant or nursing

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics
* No concurrent immunotherapy

Chemotherapy:

* See Disease Characteristics
* No concurrent chemotherapy

Endocrine therapy:

* At least 4 weeks since steroids
* No concurrent steroid therapy

Radiotherapy:

* No concurrent radiotherapy

Surgery:

* Not specified

Other:

* No concurrent immunosuppressive agents such as azathioprine or cyclosporine A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 1998-06; Primary Completion 2002-11 (Actual); Study Completion 2002-11 (Actual)

PRIMARY OUTCOMES:
Evaluate the ability of active immunotherapy with carcinoembryonic antigen (CEA) RNA pulsed dendritic cells to induce CEA specific T cells in patients with metastatic breast cancer in complete remission following peripheral blood stem cell transplant. | Following administration of 4 IV vaccine doses (1 vaccine administered every 3 weeks)

SECONDARY OUTCOMES:
Determine the clinical efficacy in terms of overall and recurrence free survival of immunotherapy with CEA RNA pulsed dendritic cells in this patients population. | Following administration of 4 IV vaccine doses (1 vaccine administered every 3 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert K. Lyerly, MD, Study Chair — Duke University
Locations (1):
- Duke Comprehensive Cancer Center, Durham, North Carolina, United States